CLINICAL TRIAL: NCT04534491
Title: An Oxytrol Transdermal System Actual Use Study (Consumer Trial of Oxytrol, Control)
Brief Title: Study to Gather Information About the Actual Use of an Adhesive Patch Placed on the Skin to Deliver Oxytrol Through the Skin Into the Bloodstream.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18165
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — oxybutynin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oxytrol (Experimental): Subjects decided to purchase Oxytrol.
  Interventions: Drug: Oxybutynin (Oxytrol, BAY839380)

INTERVENTIONS:
Drug: Oxybutynin (Oxytrol, BAY839380) — Oxybutynin transdermal patch, 3.9 mg daily (Oxytrol Transdermal System)

SUMMARY:
With this study researchers want to gather information about the consumer use behavior of Oxytrol in a simulated setting in which the medicine is sold directly to a consumer without a prescription from a healthcare professional. An area of focus was on the potential benefits of an over-the-counter status for Oxytrol and on the ongoing use behavior of the consumers. Oxytrol is a thin, flexible, clear patch that is indicated for the treatment of overactive bladder a disease characterized by a collection of symptoms, including urinary frequency, urgency, and urge incontinence. The adhesive patch is placed on the skin to deliver Oxytrol through the skin into the bloodstream.

ELIGIBILITY:
Inclusion criteria:

* Female
* 18 years of age or older
* Not pregnant or suspected to be pregnant
* Never trained or employed as a healthcare professional
* Neither the subject nor anyone in their household worked for a pharmaceutical company, a pharmacy, a managed care or health insurance company, a healthcare practice, or as a healthcare professional
* Had not participated in any market research study, product label study or clinical trial in the past 12 months

Exclusion criteria:

* Symptoms of blood in the urine not related to menses
* Back pain and fever in conjunction with frequency or urgency and any of the following: dysuria, hematuria, or cloudy urine
* Narrow-angle glaucoma
* Pregnant (as determined by a urine pregnancy test among women of child bearing potential)
* Breastfeeding
* Known allergy to oxybutynin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 855 (Actual)
Dates: Start 2010-05-25 (Actual); Primary Completion 2011-06-22 (Actual); Study Completion 2011-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Stevenson Family Pharmacy, Saint Joseph, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted in US-sites and pharmacies from 25May2010 (first patient first visit) to 22Jun2011 (last patient last visit).
Pre-assignment Details: Twelve hundred thirty (1230) women arrived at the pharmacies for the enrollment phase and 855 qualified participants purchased Oxytrol and entered the actual use phase.
Groups:
- Oxybutynin (Oxytrol, BAY839380): Subjects decided to purchase Oxytrol.
Period: Overall Study
Arm/Group | Oxybutynin (Oxytrol, BAY839380)
Started | 855
Treated | 727
Completed | 703
Not Completed | 152
Not completed — Not completed end-of-study interview | 24
Not completed — Non-users | 70
Not completed — Non-verifiable users | 58

BASELINE CHARACTERISTICS:
Arm/Group | Oxybutynin (Oxytrol, BAY839380)
Number analyzed (Participants) | 855
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: 727 verified users.
  Years
    number analyzed (Participants) | 727
    (all) | 58.4 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 727 verified users.
  Participants
    number analyzed (Participants) | 727
    Female | 727
    Male | 0
Race/Ethnicity, Customized [Number; unit: Participants] — Population: 727 verified users
  Participants
    White: number analyzed (Participants) | 727
    White | 561
    Black or African American: number analyzed (Participants) | 727
    Black or African American | 66
    Hispanic or Latino: number analyzed (Participants) | 727
    Hispanic or Latino | 64
    Asian: number analyzed (Participants) | 727
    Asian | 12
    Other: number analyzed (Participants) | 727
    Other | 24

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Who Did Not Stop Use When They Either Developed a New Symptom Referred to Anywhere in the Labeling or When Their Condition Worsened Including Abdominal and/or Pelvic Pain.
Description: For each participant who was defined as a primary endpoint misuser (i.e., subjects who did not stop using Oxytrol when they either developed a new symptom referred to anywhere in the labeling, with the addition of abdominal and/or pelvic pain, or when their OAB condition worsened) the full case report form was reviewed in order to determine if there were factors that would mitigate the incorrect decision to continue use. For example, if the subject had consulted a physician and was told to continue use, such continuation is acceptable. This process is termed "mitigation," because it involves determining if there are mitigating factors in the decision to continue use without posing any significant medical risk. Mitigation was conducted independently post-hoc by an external panel of advisors including two urologists and an urogynecologist and one physician employed by the sponsor.
Time Frame: Approximately 15 weeks from subjects' initial purchase of Oxytrol
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Oxybutynin (Oxytrol, BAY839380)
Number analyzed (Participants) | 727
Percentage of participants
  Pre-mitigation | 14.4 [12.0 to 17.2]
  Post-mitigation | 3.4 [2.2 to 5.0]

2. Secondary Outcome: The Percentage of Verified Users Who Did Not Stop Use When Their Condition Worsened or They Developed a New Symptom Referred to in the Labeling.
Description: This outcome measure did not include participants who developed abdominal and/or pelvic pain and was more reflective of how consumers stopped use according to the symptoms described on the Oxytrol labeling used in the study.
Time Frame: Approximately 15 weeks from subjects' initial purchase of Oxytrol
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Oxybutynin (Oxytrol, BAY839380)
Number analyzed (Participants) | 727
Percentage of participants
  Pre-Mitigation | 13.1 [10.7 to 15.7]
  Post-Mitigation | 3.2 [2.0 to 4.7]

3. Secondary Outcome: The Median Time Taken to Discontinue Oxytrol Use by Verified Users Who Did Not Experience Improvement in Their Symptoms After Two Weeks of Treatment.
Description: This outcome measure evaluated the number of days it took for a subject to discontinue use of Oxytrol after their symptoms worsened or had stayed the same after 2 weeks of treatment. This was calculated using diary card data.
Time Frame: Approximately 15 weeks from subjects' initial purchase of Oxytrol
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Oxybutynin (Oxytrol, BAY839380)
Number analyzed (Participants) | 187
Days | 35 [26 to 46]

4. Secondary Outcome: The Percentage of Verified Users Who Did Not Stop Oxytrol Use Within Two Weeks After Experiencing no Improvement in Their Symptoms.
Description: Factors considered in this mitigation included providing: a response to one or more open ended questions that indicated a thoughtful, informed reason for continuing use; the subject talked to a physician, and the physician advised the subject that it was acceptable to continue using product; the subject had improved by Week 7 and indicated a thoughtful, informed reason for continuing use; as well as other reasons explained in the guidelines.
  This outcome measure was analyzed based on pre- and post-mitigation assessments but the post-mitigation analysis includes all subject data and is a better reflection of the subject's overall behavior. This was calculated by dividing the total number of subjects by the number of subjects who used the Oxytrol patch at least once.
Time Frame: Approximately 15 weeks from subjects' initial purchase of Oxytrol
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Oxybutynin (Oxytrol, BAY839380)
Number analyzed (Participants) | 643
Percentage of participants
  All Subjects Pre-Mitigation | 22.6 [19.4 to 26.0]
  All Subjects Post-Mitigation | 11.0 [8.7 to 13.7]

5. Secondary Outcome: Number of Participants With Medical Risk Associated With the Development of New Symptoms or When Symptoms Did Not Improve for Patients That Continued Oxytrol Treatment.
Description: The medical risk of the newly developed symptom(s) or no sign of symptom improvement was categorized according to prospectively defined medical risk categories of 'medical risk', 'possible medical risk', and minimal/insignificant medical risk'. Mitigated data was not included in this endpoint.
Time Frame: Approximately 15 weeks from subjects' initial purchase of Oxytrol
Population: 324 participants continued Oxytrol therapy and experienced new symptoms of interest or whose OAB symptoms did not improve.
Measure: Count of Participants; unit: Participants
Arm/Group | Oxybutynin (Oxytrol, BAY839380)
Number analyzed (Participants) | 324
Participants
  Medical risk (subjects) | 16
  Possible medical risk (subjects) | 24
  Minimal/insignificant medical risk (subjects) | 284

6. Secondary Outcome: The Percentage of Verified Users Who Misused the Patch (Incorrect Duration of Use or Simultaneous Use).
Description: Factors considered in this mitigation for incorrect duration included most of the duration of patch use being correct, subject indicated understanding of the label but perhaps forgetting for a patch or two, etc. Factors considered in mitigation for simultaneous use include obvious diary errors, a subject stating that she did not do this, or a subject's doctor telling her to wear two patches at a time.
Time Frame: Approximately 15 weeks from subjects' initial purchase of Oxytrol
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Oxybutynin (Oxytrol, BAY839380)
Number analyzed (Participants) | 727
Percentage of participants
  Total Subjects Pre-Mitigation | 51.7 [47.9 to 55.4]
  Total Subjects Post-Mitigation | 21.2 [18.3 to 24.4]

ADVERSE EVENTS:
Time Frame: 15 weeks
Arm/Group | Oxybutynin (Oxytrol, BAY839380)
Serious Adverse Events (participants affected / at risk) | 35/785
Other Adverse Events (participants affected / at risk) | 509/785
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxybutynin (Oxytrol, BAY839380) (N=785)
Arrhythmia (Cardiac disorders) | 1
Cardiac disorder (Cardiac disorders) | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 2
Hepatic failure (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Pelvic inflammatory disease (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Anaesthetic complication (Injury, poisoning and procedural complications) | 1
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Schizoaffective disorder (Psychiatric disorders) | 1
Pelvic prolapse (Reproductive system and breast disorders) | 1
Uterine prolapse (Reproductive system and breast disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oxybutynin (Oxytrol, BAY839380) (N=785)
Vertigo (Ear and labyrinth disorders) | 2
Cataract (Eye disorders) | 5
Dry eye (Eye disorders) | 10
Vision blurred (Eye disorders) | 5
Visual acuity reduced (Eye disorders) | 3
Visual impairment (Eye disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal pain lower (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 20
Diarrhoea (Gastrointestinal disorders) | 16
Dry mouth (Gastrointestinal disorders) | 32
Faecal incontinence (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 16
Toothache (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Application site erythema (General disorders) | 9
Application site irritation (General disorders) | 142
Application site pruritus (General disorders) | 8
Application site rash (General disorders) | 4
Application site reaction (General disorders) | 13
Fatigue (General disorders) | 11
Irritability (General disorders) | 3
Oedema peripheral (General disorders) | 4
Hypersensitivity (Immune system disorders) | 7
Seasonal allergy (Immune system disorders) | 3
Bronchitis (Infections and infestations) | 10
Cystitis (Infections and infestations) | 16
Diverticulitis (Infections and infestations) | 3
Fungal infection (Infections and infestations) | 6
Gastroenteritis viral (Infections and infestations) | 8
Herpes zoster (Infections and infestations) | 2
Infection (Infections and infestations) | 2
Influenza (Infections and infestations) | 18
Nasopharyngitis (Infections and infestations) | 46
Pharyngitis streptococcal (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 21
Tooth infection (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 47
Vulvovaginal mycotic infection (Infections and infestations) | 2
Arthropod bite (Injury, poisoning and procedural complications) | 2
Contusion (Injury, poisoning and procedural complications) | 2
Excoriation (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 3
Joint sprain (Injury, poisoning and procedural complications) | 3
Skin laceration (Injury, poisoning and procedural complications) | 3
Wrist fracture (Injury, poisoning and procedural complications) | 3
Blood cholesterol increased (Investigations) | 4
Blood glucose increased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 17
Flank pain (Musculoskeletal and connective tissue disorders) | 4
Joint swelling (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Osteopenia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 2
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Balance disorder (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 15
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 20
Migraine (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Sciatica (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 14
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 3
Dysuria (Renal and urinary disorders) | 12
Haematuria (Renal and urinary disorders) | 3
Hypertonic bladder (Renal and urinary disorders) | 5
Micturition urgency (Renal and urinary disorders) | 4
Urge incontinence (Renal and urinary disorders) | 24
Urinary incontinence (Renal and urinary disorders) | 3
Urinary retention (Renal and urinary disorders) | 7
Urine odour abnormal (Renal and urinary disorders) | 5
Breast tenderness (Reproductive system and breast disorders) | 2
Menorrhagia (Reproductive system and breast disorders) | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Dry throat (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Blister (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Hot flush (Vascular disorders) | 2
Hypertension (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days